CLINICAL TRIAL: NCT07339657
Title: Evaluation of the Validity and Reliability of the Protection, Amount, Frequency, Compliance, Body Image (PRAFAB) Questionnaire in Women With Urinary Incontinence
Brief Title: Validity and Reliability of the PRAFAB
Status: Recruiting | Type: Observational
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Emel Taşvuran Horata, PhD; Associate Professor, Afyonkarahisar Health Sciences University
Other Study IDs: 291
Record Dates: First submitted 2026-01-05; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Urinary Incontinence
Keywords: urinary incontinence; validity; reliability
MeSH Terms: conditions — Urinary Incontinence | interventions — Reproducibility of Results

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Urinary Incontinence: All subtypes of urinary incontinence (stress urinary incontinence, urge incontinence, etc.) were included in our study.
  Interventions: Other: Construct validity; Other: Test-retest reliability

INTERVENTIONS:
Other: Construct validity — This is not an intervention. This is an analysis conducted to examine the factor structure of this questionnaire. The analysis will be performed using the SPSS 26.0 software package program.
  Other Names: Exploratory Factor Analysis
Other: Test-retest reliability — This is not an intervention. This is an analysis conducted to examine the repeatability of this questionnaire. The analysis will be performed using the SPSS 26.0 software package program.

SUMMARY:
PRAFAB assesses both the objective and subjective aspects of urinary incontinence. While differing from other questionnaires in this respect, it consists of only five questions. Today, there is a need for multidimensional and easy-to-use scales that can assess the effects of incontinence on quality of life. Therefore, the aim of this study is to conduct a Turkish validity and reliability study of the PRAFAB questionnaire in women with urinary incontinence.

DETAILED DESCRIPTION:
PRAFAB assesses both the objective and subjective aspects of urinary incontinence. While differing from other questionnaires in this respect, it consists of only five questions. Today, there is a need for multidimensional and easy-to-use scales that can assess the effects of incontinence on quality of life. Therefore, the aim of this study is to conduct a Turkish validity and reliability study of the PRAFAB questionnaire in women with urinary incontinence.

In this context, the study consists of two phases. In the first phase, the PRAFAB questionnaire was translated into Turkish and culturally adapted; in the second phase, the validity and reliability analyses of the Turkish version of the PRAFAB questionnaire (PRAFAB-Turkish) were conducted.

The study will be conducted by Afyonkarahisar University of Health Sciences. Participants consisted of women who presented as outpatients at the AFSU Health Application and Research Center Urology Clinic and were diagnosed with urinary incontinence by a urologist.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older
* Have been diagnosed with urinary incontinence by a urologist
* Be female

Exclusion Criteria:

* Being pregnant,
* Being in the early postpartum period,
* Have been diagnosed with bladder cancer, diabetic nephropathy, a history of central nervous system damage, congenital urological disorders, urinary tract infection, neurogenic bladder, severe cognitive impairment, and severe psychiatric illness.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants aged 18 years and older with female urinary incontinence will be included in the study. Participants will consist of women who visit the AFSU Health Application and Research Center Urology Outpatient Clinic and are diagnosed with urinary incontinence by a urologist.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
PRAFAB | This questionnaire, which takes approximately 2-3 minutes to complete, will be administered to participants twice at two-week intervals.
  It is a 5-item questionnaire. Developed to assess the severity of urinary incontinence and its impact on the individual.

CONTACTS AND LOCATIONS:
Overall Officials: EMEL TAŞVURAN HORATA, Principal Investigator — Afyonkarahisar Sağlık Bİlimleri Üniversitesi; Şeyma Betül İNCE, Study Chair — No Affiliation; Harun TAŞKIN, PhD, Study Chair — Afyonkarahisar Health Sciences University; Osman GERÇEK, MD, Study Chair — Afyonkarahisar Health Sciences University; Mustafa Esat İNCE, MD, Study Chair — Afyonkarahisar Health Sciences University; Bary Berghmans, Assoc. Prof., Study Chair — Maastricht University
Locations (1):
- Emel Taşvuran Horata, Afyonkarahisar, Merkez, Turkey (Türkiye)